CLINICAL TRIAL: NCT01047163
Title: Maintenance of Muscle Mass in Older People: the Negative Impact of Statin Therapy
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RB03DR
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Myopathy
Keywords: Muscle soreness; Simvastatin; Men; Muscle Atrophy
MeSH Terms: conditions — Muscular Diseases; Myalgia; Multiple Endocrine Neoplasia Type 1; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Muscle biopsy, Serum & Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Statin: Men aged 65-75yr on Simvastatin therapy presenting with muscle soreness
- Control: Men, aged 65-75yr not on Statin therapy

SUMMARY:
A major contributor to frailty and immobility in the elderly is the age related loss of muscle mass (sarcopenia). Cardiovascular disease (CVD) is the leading cause of mortality in the elderly, with high blood cholesterol and lipids being the major modifiable risk factor. Statins reduce blood cholesterol, but muscle related pain, tenderness and discomfort (myopathy) is an adverse event associated with statin therapy, with older people being at a much greater risk. Statin myopathy presents as muscle aches and weakness, with or without evidence of muscle damage; however the underlying mechanisms responsible for these symptoms are poorly understood. Using an animal model, the applicants have shown the main pathway regulating muscle protein synthesis is inhibited in statin myopathy, and genes regulating muscle protein breakdown, the inhibition of muscle carbohydrate use and inflammation are dramatically increased. Therefore we wish to determine whether these changes are seen in the muscle of older people with symptoms of statin myopathy, and whether this is associated with lower muscle mass and impaired muscle function compared with older people with no history of statin use. Identification of the mechanisms involved in statin myopathy could lead to effective therapy for older people unable to tolerate statins.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality in elderly people accounting for >208,000 deaths each year, with hyperlipidaemia being the major modifiable risk factor in the elderly. Statins inhibit synthesis of cholesterol, and their therapy has been associated with a 30% reduction in cardiovascular events. Statins are generally well tolerated, but can have myopathic effects. Randomised trials suggest rhabdomyolysis (> 10 times the upper limit of normal serum creatine kinase (CK)) is rare, and even myalgia and myositis (muscle aches or weaknesses with and without increases in serum CK, respectively), although more common, are not highly prevalent. However, the incidence of adverse muscular events associated with the most commonly prescribed statin, simvastatin, is high, particularly at high doses (18%), and given the recommendation by National Institute for Health and Care Excellence to prescribe simvastatin over other statins, adverse muscular events could potentially increase further with increased use, and particularly in the elderly who are at a far greater risk [1]. Using an animal model, the applicants have shown that the principal pathway thought to regulate muscle protein synthesis (the phosphatidylinositol 3-kinase/Protein Kinase B (PI3k/Akt) signalling pathway) is down regulated in simvastatin induced myopathy [2]. Furthermore, this was paralleled by the marked up regulation of genes thought to increase muscle protein breakdown, impair carbohydrate oxidation, and increase oxidative stress and inflammation. We will test the hypotheses: (i) That people over 65 years of age prescribed simvastatin, and experiencing muscle related aches and pains, will present with exacerbated muscle mass loss and impaired muscle function (strength and fatigability) compared to age and sex matched control volunteers (statin free). (ii) That signaling pathways and genes seen to be dysregulated in an animal model of simvastatin induced myopathy will also be dysregulated in the muscle of older people prescribed simvastatin and experiencing muscle related aches and pains, and may thereby underpin the symptoms associated with statin myopathy. We will recruit 15, male volunteers > 65 years of age reporting myopathic symptoms with simvastatin administration and 15 age and sex matched control volunteers (statin free). Volunteers will be deemed suitable for entry into a statin myopathy group if they show elevated serum CK, muscle tenderness, reduced isometric strength [for their age] and appropriate scoring of a muscle pain questionnaire. All volunteers will undertake two experimental visits: Visit 1 to determine body composition, muscle strength and fatigability, and Visit 2 to undergo an insulin clamp lasting 3 hours. Visit 1 will involve measurement of body composition using dual energy X-ray absorptiometry (DEXA), and isometric strength and fatigability of the knee extensor muscles using an exercise dynamometer. Visit 2 will involve muscle protein synthesis, leg protein breakdown and glucose disposal being determined, using a primed constant infusion of stable isotope labeled amino acids during a two-stage 180 min insulin clamp at rest (see detailed protocol for specifics). In short, a basal muscle biopsy will be obtained (Vastus lateralis), after which serum insulin will be clamped at the fasted concentration (~5 mU/l) for the first 90 min, allowing processes that govern protein breakdown to occur without any inhibitory effect of raised serum insulin, and will be followed by a second muscle biopsy. For the remaining 90 min, serum insulin will be raised equivalent to the fed state by the administration of 30 milliunit (mU).m-2.min-1 insulin, along with a variable infusion of 20% glucose to maintain plasma glucose concentration at 4.5 mmol.l-1. Also a constant infusion of mixed amino acids will be administered (10g per hour) allowing protein synthesis to be examined. Furthermore, insulin resistance will be estimated during this second 90 min by measuring leg glucose disposal. A third muscle biopsy sample will be obtained after this second 90 min period of investigation. Determination of muscle protein synthesis and leg protein breakdown will necessitate a femoral vein catheter being inserted for venous blood sampling, a cannula being inserted retrograde into a superficial vein of a heated hand for sampling of arterialised-venous blood, and a cannula being placed in the antecubital vein of both forearms for the infusion of mixed amino acids, as well as octreotide, glucose and insulin. Femoral arterial and femoral venous blood flow will be determined using Doppler ultrasound, which is completely non-invasive. Body composition and leg isometric strength and fatigue will be determined (Visit 1). Muscle biopsy samples and blood samples will be used to determine rates of muscle protein synthesis, breakdown and glucose disposal. Muscle biopsy samples will also be used to examine the expression of genes and proteins that regulate muscle protein balance, inflammation and carbohydrate metabolism. Sample size is based on the observed increase in atrophy gene (MAFbx) expression in muscle of statin treated individuals [3]. A 2 fold increase in MAFbx messenger ribonucleic acid (mRNA) (standard deviation = 0.3 fold) was reported in muscle from 8 individuals treated with statins experiencing myopathic symptoms compared to controls. Therefore, assuming a power of 80%, 7 subjects would be required to detect an effect. Being conservative, and accounting for some drop outs, we will recruit 15 volunteers per group to ensure sufficient statistical power. There are currently no measures of muscle protein synthesis, degradation or anabolic signaling proteins in people reporting statin myopathy on which to base additional power calculations, but studies in people between 65-85 years of age in which such measurements have been made by the applicants have involved similar numbers of men and women.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 65-75yrs
* Simvastatin use with muscle soreness or no statin use
* Residing in Nottinghamshire area

Exclusion Criteria:

* Clotting disorders or previous Cerebral Vascular Accident /Transient Ischaemic Attack /Deep Vein Thrombosis
* Metabolic disease e.g. diabetes, thyroid dysfunction
* Inflammatory conditions e.g. Rheumatoid Arthritis, Crohn's Disease
* Tobacco smoker
* Lower limb circulation problems e.g. Claudication
* Epilepsy
* Renal pathology
* Respiratory problems including Asthma

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase in MAFbx (atrophy gene) mRNA expression in those on Statin therapy | On study visit

SECONDARY OUTCOMES:
Expression of genes that regulate muscle protein balance. | Before, 2 hours after aminoacid tracer infusion and 2 hours after a 40 mU/m2 hyperinsulinaemic, euglycaemic clamp with aminoacid infusion (10g/h)

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Greenhaff, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Physiology Laboratories, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nichols GA, Koro CE. Does statin therapy initiation increase the risk for myopathy? An observational study of 32,225 diabetic and nondiabetic patients. Clin Ther. 2007 Aug;29(8):1761-70. doi: 10.1016/j.clinthera.2007.08.022. PMID 17919557
- [Background] Mallinson JE, Constantin-Teodosiu D, Sidaway J, Westwood FR, Greenhaff PL. Blunted Akt/FOXO signalling and activation of genes controlling atrophy and fuel use in statin myopathy. J Physiol. 2009 Jan 15;587(1):219-30. doi: 10.1113/jphysiol.2008.164699. Epub 2008 Nov 10. PMID 19001041
- [Background] Hanai J, Cao P, Tanksale P, Imamura S, Koshimizu E, Zhao J, Kishi S, Yamashita M, Phillips PS, Sukhatme VP, Lecker SH. The muscle-specific ubiquitin ligase atrogin-1/MAFbx mediates statin-induced muscle toxicity. J Clin Invest. 2007 Dec;117(12):3940-51. doi: 10.1172/JCI32741. PMID 17992259
- [Result] Mallinson JE, Marimuthu K, Murton A, Selby A, Smith K, Constantin-Teodosiu D, Rennie MJ, Greenhaff PL. Statin myalgia is not associated with reduced muscle strength, mass or protein turnover in older male volunteers, but is allied with a slowing of time to peak power output, insulin resistance and differential muscle mRNA expression. J Physiol. 2015 Mar 1;593(5):1239-57. doi: 10.1113/jphysiol.2014.285577. Epub 2015 Jan 26. PMID 25620655